CLINICAL TRIAL: NCT02156401
Title: VTEval Project - Three Observational, Prospective Cohort Studies Including Biobanking to Evaluate and Improve Diagnostics, Management Strategies and Risk Stratification in Venous Thromboembolism
Brief Title: VTEval Project - Prospective Cohort Studies to Evaluate and Improve Diagnostics, Management Strategies and Risk Stratification in VTE
Acronym: VTEval
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Maastricht University (Other); Hochschule Fresenius (Other); University of Bonn (Other); Siemens Corporation, Corporate Technology (Industry); Bayer (Industry); Eurofins (Industry)
Responsible Party: Principal Investigator, Philipp Wild, MD, MSc, Univ.-Prof. Dr. med. Philipp Wild, MSc, Johannes Gutenberg University Mainz
Other Study IDs: UMCM-2013EPI02
Record Dates: First submitted 2014-05-23; First posted 2014-06-05 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Venous Thromboembolism (VTE); Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE)
Keywords: Venous thromboembolism; Deep vein thrombosis; Pulmonary embolism; Cohort study/epidemiology; Outcome; Prognosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Na-Citrated Plasma, EDTA-Plasma, DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Suspect of Pulmonary Embolism (PE)
- Cohort 2: Suspect of Deep Vein Thrombosis (DVT)
- Cohort 3: Incidental Venous Thromboembolism (VTE)

SUMMARY:
Venous thromboembolism (VTE) with its two clinical manifestations deep vein thrombosis (DVT) and pulmonary embolism (PE) is a life-threatening disease that is associated with considerable morbidity and mortality. The incidence of VTE increases with age and it - as the third most common cardiovascular disease after ischemic heart disease and stroke - represents an important public health problem in industrialized countries with several aspects in need to be addressed.

VTEval Project includes three long-term prospective observational studies to evaluate and improve VTE diagnostics and management, treatment and outcome. The aims of the project include a systematic assessment of VTE, i.e. disease status (symptoms, clinical and subclinical aspects) and risk profiles (classic, psychosocial and environmental factors), using a system-oriented approach. VTEval collects three large prospective cohorts of patients with suspected and incident VTE consisting of individuals with a clinical suspicion of acute PE, individuals with a clinical suspicion of acute DVT, and individuals with incidental diagnosis of VTE).

The standardized and harmonized data acquisition of the study establishes a sustainable resource for comprehensive research on VTE, thus providing the basis for both short- and long-term analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and Informed written consent
* Clinical condition:

  * Cohort 1: Clinical suspicion of acute PE (with or without DVT)
  * Cohort 2: Clinical suspicion of acute DVT (without symptomatic PE)
  * Cohort 3: Incidentally diagnosed VTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals either with clinically suspected or incident diagnosis of VTE
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | Baseline
  Overall mortality, consisting of:
  * PE-related death
  * All other causes of death
Symptomatic venous thromboembolism | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
  Composed by:
  * PE-related death
  * Development or recurrence of nonfatal PE
  * Development or recurrence of DVT

SECONDARY OUTCOMES:
Hemodynamic instability | Baseline
  Defined as at least one of the following:
  * Cardiopulmonary resuscitation (CPR) or defibrillation
  * Cardiogenic shock or need of catecholamine administration
  * Systolic blood pressure < 90mm Hg, or a pressure drop by more than 40mm Hg for >15 min
Use of mechanical ventilation | Baseline
Admission to Intensive Care Unit (ICU) | Baseline
Recurrence of acute PE | Baseline
Cardiac dysfunction or heart failure | Baseline
Pneumonia | Baseline
Symptomatic and/or asymptomatic DVT | Baseline
Major bleeding | Baseline
Clinically relevant non-major bleedings | Baseline
Diagnostic of a previously unknown malignancy | Baseline
Length of hospitalization | Baseline
Implantation of vena cava filter | Baseline
Thrombolytic treatment | Baseline
Interventional treatment | Baseline
Surgery | Baseline
Overall mortality | Assessment at month 3/6 and 12; year 2-6 (Active follow-up)
PE-related death | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Development or recurrence of clinical symptomatic PE/DVT | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Asymptomatic DVT | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Chronic venous insufficiency (CVI) | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Post-thrombotic Syndrome (PTS) | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Development of cardiac dysfunction or heart failure | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Development of pulmonary hypertension | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Respiratory dysfunction | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Major bleeding | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Clinically relevant non-major bleedings | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Diagnostic of a previously unknown malignancy | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Net clinical outcome (NCO) | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
O2 home treatment | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Pulmonary vasoactive drugs | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Development of Chronic Thromboembolic Pulmonary Hypertension (CTEPH) | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Hospitalization | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Length of stay in Hospital due to VTE | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Major adverse cardiac and cerebrovascular event (MACCE) | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Cardiovascular event | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)
Cerebrovascular event | Assessment at month 3, 6 and 12; year 2-6 (Active follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp S Wild, MD, MSc, Principal Investigator — University Medical Center of Johannes Gutenberg University Mainz, Germany
Locations (1):
- University Medical Center of the Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Ten Cate V, Eggebrecht L, Schulz A, Panova-Noeva M, Lenz M, Koeck T, Rapp S, Arnold N, Lackner KJ, Konstantinides S, Espinola-Klein C, Munzel T, Prochaska JH, Wild PS. Isolated Pulmonary Embolism Is Associated With a High Risk of Arterial Thrombotic Disease: Results From the VTEval Study. Chest. 2020 Jul;158(1):341-349. doi: 10.1016/j.chest.2020.01.055. Epub 2020 Mar 23. PMID 32217063
- [Derived] Frank B, Ariza L, Lamparter H, Grossmann V, Prochaska JH, Ullmann A, Kindler F, Weisser G, Walter U, Lackner KJ, Espinola-Klein C, Munzel T, Konstantinides SV, Wild PS; VTEval study group. Rationale and design of three observational, prospective cohort studies including biobanking to evaluate and improve diagnostics, management strategies and risk stratification in venous thromboembolism: the VTEval Project. BMJ Open. 2015 Jul 1;5(7):e008157. doi: 10.1136/bmjopen-2015-008157. PMID 26133379